CLINICAL TRIAL: NCT06037057
Title: Application of Artificial Intelligence Deep Learning Technology in Magnetic Resonance Lumbar Imaging
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LY2023-121-B
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Deep Learning,Lumbar Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention name — no intervention description

SUMMARY:
To study the comparative analysis of artificial intelligence deep learning technology in the image quality of under-artificial intelligence (AI) reconstruction images and the original acquisition images of magnetic resonance lumbar spine

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged ≥18 years, with no history of lumbar surgery, underwent lumbar magnetic resonance imaging examination.

Exclusion Criteria:

* With metal implants in the body, claustrophobic, unable to lie flat for 15 minutes, with a history of lumbar surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of both sexes, aged ≥18 years, with no history of lumbar surgery, underwent lumbar magnetic resonance imaging examination.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-08 (Estimated); Primary Completion 2024-03-08 (Estimated); Study Completion 2024-03-08 (Estimated)

PRIMARY OUTCOMES:
Application of Artificial Intelligence Deep Learning Technology in Magnetic Resonance Lumbar Imaging | 2025.3-2025.6
  manuscript